CLINICAL TRIAL: NCT07246525
Title: Cluster Randomized Trial of Intermittent Preventive Treatment of Malaria in School-age Children to Improve the Health of Students and Decrease Community Transmission
Brief Title: Intermittent Preventive Treatment of Malaria in School-age Children to Decrease Community Transmission
Acronym: CRITICal
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Infectious Diseases Research Collaboration, Uganda (Other); Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRITICal; U01AI186861 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Malaria
Keywords: intermittent preventive treatment; school children; dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: This study will be an open label, phase IV, cluster-randomized trial to evaluate the effectiveness of IPTsc with DP administered approximately every 2 months to children attending primary school. Clusters are geographically defined target areas surrounding government-run health facilities previously established and referred to as Malaria Reference Centers (MRCs). A total of 24 clusters (MRCs) will be included in the study. These clusters were selected based on participation in an on-going sentinel site malaria surveillance network in areas with moderate-high malaria transmission intensity. Clusters will be randomized in a 1:1 ratio such that all primary schools serving the populations of each target area will either receive IPTsc or not receive IPTsc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPTsc (Experimental): DP will be administered approximately every 2 months for two years to all eligible children enrolled in primary schools serving the target areas from clusters randomized to the interventional arm.
  Interventions: Drug: dihydroartemisinin-piperaquine
- No IPTsc (No Intervention): No IPTsc (standard of care)

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — D-Artepp, is manufactured by Guilin Pharmaceutical Co Ltd, and is prequalified by the WHO and approved for use in Uganda by the National Drug Authority. Standard treatment doses of DP (once a day x 3 days) will be administered using weight-based guidelines targeting a total dose of 6.4 mg/kg dihydroartemisinin and 51.2 mg/kg of piperaquine as per manufacturer's instructions.
  Other Names: D-Artepp
  Arms: IPTsc

SUMMARY:
The CRITICal study aims to estimate the effectiveness of intermittent preventive treatment in school children (IPTsc) with dihydroartemisinin-piperaquine (DP) for reducing community level malaria burden. Given that school-aged children are the primary drivers of transmission, the study hypothesis is that IPTsc will reduce this infectious reservoir and thus the burden of malaria in persons of all ages in surrounding communities.

DETAILED DESCRIPTION:
The CRITICal study is an open label, phase IV, cluster-randomized trial to evaluate the effectiveness of IPTsc with DP administered approximately every 2 months to children attending primary school. Clusters are geographically defined target areas surrounding government-run health facilities previously established and referred to as Malaria Reference Centers (MRCs). A total of 24 clusters (MRCs) will be included in the study. These clusters were selected based on participation in an on-going sentinel site malaria surveillance network in areas with moderate-high malaria transmission intensity. Clusters will be randomized in a 1:1 ratio such that all primary schools serving the populations of each target area will either receive IPTsc or not receive IPTsc. The intervention will be delivered for 2 years and evaluations will continue for 1 additional year after the intervention is stopped. The primary outcome of the study will be malaria incidence within the population of the target areas. Secondary outcomes will include the the prevalence of parasitemia and molecular markers of DP resistance at the community level; the prevalence of parasitemia, anemia, and school attendance among children attending primary school; and estimates of the cost-effectiveness of IPTsc.

ELIGIBILITY:
Inclusion Criteria:

* Child currently attending the participating school.
* Agreement of parent/guardian to provide informed consent.
* Agreement of children aged 8-17 years to provide assent.

Exclusion Criteria:

* Missing school on three consecutive days of the school survey.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4800 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of cases of laboratory-confirmed malaria diagnosed among patients residing in the target area during the period the intervention is implemented | 24 months after intervention implemented
  malaria incidence: the number of cases of laboratory-confirmed malaria diagnosed at the MRC among patients residing in the target area, per unit time, divided by the total population of the target area in patients of all ages over the 24-month intervention period

SECONDARY OUTCOMES:
Number of cases of laboratory-confirmed malaria diagnosed among patients residing in the target area after the intervention is competed | 12 months after intervention is completed
  malaria incidence: the number of cases of laboratory-confirmed malaria diagnosed at the MRC among patients residing in the target area, per unit time, divided by the total population of the target area in patients of all ages 12 months after intervention is completed
Parasite prevalence among community residents 12 months after the intervention is implemented | 12 months after the intervention is implemented
  Proportion of blood smears positive for parasites by microscopy at the time of community cross-sectional surveys
Parasite prevalence among community residents 24 months after the intervention is implemented | 24 months after the intervention is implemented
  Proportion of blood smears positive for parasites by microscopy at the time of community cross-sectional surveys
Parasite prevalence among community residents 12 months after the intervention is completed | 12 months after the intervention is completed
  Proportion of blood smears positive for parasites by microscopy at the time of community cross-sectional surveys
Prevalence of molecular markers of DP resistance from parasite positive samples from community surveys 12 months after the intervention is implemented | 12 months after the intervention is implemented
  Proportion of parasite positive samples with molecular markers of DP resistance detected
Prevalence of molecular markers of DP resistance from parasite positive samples from community surveys 24 months after the intervention is implemented | 24 months after the intervention is implemented
  Proportion of parasite positive samples with molecular markers of DP resistance detected
Prevalence of molecular markers of DP resistance from parasite positive samples from community surveys 12 months after the intervention is completed | 12 months after the intervention is completed
  Proportion of parasite positive samples with molecular markers of DP resistance detected
Parasite prevalence among schoolchildren 12 months after the intervention is implemented | 12 months after the intervention is implemented
  Proportion of blood smears positive for parasites by microscopy at the time of school surveys
Parasite prevalence among schoolchildren 24 months after the intervention is implemented | 24 months after the intervention is implemented
  Proportion of blood smears positive for parasites by microscopy at the time of school surveys
Parasite prevalence among schoolchildren 12 months after the intervention is completed | 12 months after the intervention is completed
  Proportion of blood smears positive for parasites by microscopy at the time of school surveys
Anemia prevalence among schoolchildren 12 months after the intervention is implemented | 12 months after the intervention is implemented
  Proportion of children with anemia at the time of school surveys
  Anemia defined based on WHO criteria as:
  1. hemoglobin less than 11.5g/dl in children 5 - 11 years of age;
  2. hemoglobin less than 12.0g/dl in children 12 - 14 years of age and non-pregnant girls 15 years and above; and
  3. hemoglobin less than 13.0g/dl in boys 15 years and above) 12 and 24 months after the intervention is implemented and school attendance (defined as the number of days attending school / number of days school in session) over the 24-month intervention period
Anemia prevalence among schoolchildren 24 months after the intervention is implemented | 24 months after the intervention is implemented
  Proportion of children with anemia at the time of school surveys
  Anemia defined based on WHO criteria as:
  1. hemoglobin less than 11.5g/dl in children 5 - 11 years of age;
  2. hemoglobin less than 12.0g/dl in children 12 - 14 years of age and non-pregnant girls 15 years and above; and
  3. hemoglobin less than 13.0g/dl in boys 15 years and above) 12 and 24 months after the intervention is implemented and school attendance (defined as the number of days attending school / number of days school in session) over the 24-month intervention period
Anemia prevalence among schoolchildren 12 months after the intervention is completed | 12 months after the intervention is completed
  Proportion of children with anemia at the time of school surveys
  Anemia defined based on WHO criteria as:
  1. hemoglobin less than 11.5g/dl in children 5 - 11 years of age;
  2. hemoglobin less than 12.0g/dl in children 12 - 14 years of age and non-pregnant girls 15 years and above; and
  3. hemoglobin less than 13.0g/dl in boys 15 years and above) 12 and 24 months after the intervention is implemented and school attendance (defined as the number of days attending school / number of days school in session) over the 24-month intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No